CLINICAL TRIAL: NCT04359082
Title: The Effects of Cocoa-rich Bioflavanol Supplementation on Manual Dexterity During Cold Exposure
Brief Title: Cocoa-rich Bioflavanol Supplementation Effects During Cold Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-27-H
Record Dates: First submitted 2020-03-09; First posted 2020-04-24 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cold Exposure; Manual Dexterity; Gut Microbiome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over controlled trial
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for 8 straight days
  Interventions: Other: Placebo Pill
- Bioflavanol (Experimental): Bioflavanol supplementation for 8 days at 900 mg flavanol per day
  Interventions: Dietary Supplement: CocoaVia supplement

INTERVENTIONS:
Dietary Supplement: CocoaVia supplement — CocoaVia is a dietary supplement that has concentrated bioflavanols of 225 mg flavanols per pill along with 30 mg theobromine and 10 mg caffeine
  Arms: Bioflavanol
Other: Placebo Pill — Placebo pill has no bioflavanols with 30 mg theobromine and 10 mg caffeine
  Arms: Placebo

SUMMARY:
The primary purpose is to test whether cocoa-rich bioflavanols can improve blood flow to the hand and fingers and improve hand function/dexterity during cold exposure. Secondary purpose is to understand whether bioflavanol supplementation can change the gut microbiome.

DETAILED DESCRIPTION:
Loss of manual dexterity significantly impacts Warfighter effectiveness and lethality on the cold-weather battlefield. Identifying countermeasures that improve hand and finger temperatures, hand and finger blood flow, manual dexterity, and thermal comfort may lead to better Warfighter performance. A primary purpose of this study is to test the efficacy of a commercial off-the-shelf cocoa-rich bioflavanol product on hand/finger blood flow and temperature, manual dexterity, and thermal comfort during whole-body cold exposure. Another primary purpose is to determine the effect of bioflavanols on the finger cold-induced vasodilation (CIVD) response to cold-water immersion. Secondary purposes are to determine if: a) cocoa-rich flavanols stimulate the growth of beneficial gut bacteria and b) impact attention and effort perception during dexterity task completion in the cold. Two experimental studies (n = 20 in each study, 10 women and 10 men, 18-49 yr) will be conducted. Experiment #1 consists of immersing the middle finger in cold water (4°C) for 30 minutes; experiment #2 consists of whole-body cold exposure (8°C air, 90-min exposure, wearing cold-weather clothing but bare-handed). In both experiments, outcomes will be measured after both acute flavanol or placebo ingestion and chronic ingestion of flavanol/placebo (8 days of supplementation). Daily flavanol ingestion will be 900 mg/day. Volunteers will serve as their own controls in this crossover, double-blind research design. The washout period between flavanol and placebo treatments will be at least 2 weeks (longer for women who will be tested only during the follicular phase). Measurements during these tests include skin temperature, skin blood flow, fine and gross motor dexterity, thermal comfort, and effort perception. Fecal samples, in both experiments, will be collected before and after 8 days of cocoa-rich bioflavanol supplementation to examine if bioflavanol supplementation increases the number of beneficial bacteria in the gut microbiome. Information from this study will inform combat nutrition developers about the efficacy of cocoa-rich bioflavanols and possible inclusion into cold-weather field rations.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18-49 years (17-49 for active military).
* Refrain from the following for 2 weeks before and during the study (including the washout period): consumption of flavanol rich foods including cocoa, chocolate, apples, red, white, and sweet wine, apricots, blueberries, peaches/nectarines, plums, grapes, strawberries, pecans (no more than ½ cup/day, pistachios, (no more than ½ cup per day), and apple juice.
* Participants not to change their daily intakes of tea (green or black) or coffee.

Exclusion Criteria:

* History of cold injuries.
* Raynaud's syndrome.
* Cold-induced asthma/bronchospasm
* Difficulty swallowing pills.
* Previous hand/finger injuries that impair dexterity and hand function.
* Metal hardware (plates/screws) in the forearms and hands.
* Blood donation in last 8 weeks.
* Medicine use (including any over the counter medication such as Tylenol, Advil, Sudafed, etc…), with the exception of birth control and a multi-vitamin.
* Known allergies to medical adhesives or cocoa/chocolate.
* History of disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis; or previous gastrointestinal surgery.
* No planned MRI during the study or within 2 days after completing a cold test.
* Use of dietary supplements (to include probiotics and prebiotics), with exception of multi-vitamin containing up to 100% of the recommended daily allowance (RDA).
* No exercise or smoking within 8 hours of testing.
* Pregnant or breastfeeding.
* Oral antibiotic use within 3 months of study participation.
* Inability or unwillingness to not consume fermented food products or prebiotic-containing food products for 2 weeks prior to and throughout study participation. Examples include kefir, kombucha, aged cheese, pickles, sauerkraut, sour cream, tempeh, yogurt, kimchi, miso, vinegar, sourdough bread, wine and beer.
* Colonoscopy within 3 months of study participation.
* On average has a bowel movement less frequently than every other day.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Cold induced vasodilation response | 30 minutes
  Skin/finger temperature changes during finger immersion in 4°C water
Manual dexterity-PP | 2 hours
  Purdue Pegboard score during 8°C air exposure. Score is the number of pegs placed into board.
Manual dexterity-MRM | 2 hours
  Minnesota Rate of Manipulation dexterity score during 8°C air exposure. Score is the number of pieces put together during times period.
Hand and finger temperatures | 2 hours
  Hand and finger temperatures during cold air exposure in 8

SECONDARY OUTCOMES:
Gut microbiome | 8 days
  How do targeted populations (Bifidobacterium spp., Lactobacillus spp., C. coccoides-Eubacterium rectale, Faecalibacterium prausnitzii, Prevotella/Bacteroides, Roseburia, and Akkermansia muciniphila) change as a result of bioflavanol supplementation

CONTACTS AND LOCATIONS:
Overall Officials: John W Castellani, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- John W Castellani, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alba BK, Greenfield AM, Yurkevicius BR, Jones ML, Castellani JW. Short-term cocoa bioflavanol supplementation does not improve cold-induced vasodilation in young healthy adults. Eur J Appl Physiol. 2024 May;124(5):1523-1534. doi: 10.1007/s00421-023-05380-4. Epub 2023 Dec 27. PMID 38150009

DOCUMENTS (2):
  • Informed Consent Form: CIVD (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT04359082/ICF_000.pdf
  • Informed Consent Form: Cold Air (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT04359082/ICF_001.pdf